CLINICAL TRIAL: NCT01258569
Title: Entereg Laparoscopic Colon Resection Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hartford Hospital (Other)
Collaborators: Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JOHN002914HE
Record Dates: First submitted 2010-12-09; First posted 2010-12-13 (Estimated); Last update posted 2015-08-26 (Estimated); Status verified 2015-08

CONDITIONS: Laparoscopic Colonic Resection
Keywords: laparoscopic; colon; resection; Entereg
MeSH Terms: interventions — alvimopan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Entereg (Active Comparator)
  Interventions: Drug: Entereg
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Entereg — Alvimopan (Entereg), an oral peripherally- acting mu-opioid receptor antagonist, is the first and only drug approved by the FDA to accelerate the time to upper and lower GI recovery in after partial large or small bowel resection surgery with primary anastomosis.
  Arms: Entereg
Drug: Entereg — oral, 12 mg 30-300 min pre-op then BID up to 7 days (or 15 total doses)
  Arms: Entereg
Drug: placebo — 12 mg oral 30-300 min pre-op then BID up to 7 days (or 15 doses)
  Arms: Placebo

SUMMARY:
Entereg (Alvimopan) is a peripherally acting mu-opioid receptor antagonist that has been shown to increase postoperative bowel function in patients after open bowel resection surgery. It has been proven safe and effective for short-term in-house treatment. At the present there are several Drug Use Utilization Evaluation studies reporting results involving the use of alvimopan (ENTEREG) in laparoscopic bowel resection patients. However, this study will be the first randomized, prospective, double-blind, placebo-controlled trial looking at this population. We propose that Entereg will decrease the length of stay by one day in the laparoscopic colon resection patient. We wish to perform a voluntary, double-blinded, placebo controlled study. We plan an enrollment population of 250 patients. Twelve milligrams of Entereg will be administered 30 minutes to 5 hours pre-op followed by 12 mg BID, up to 7 days or 15 total doses. The primary endpoint of the study will be length of stay. The time of GI-2 recovery (toleration of solid food and first bowel movement) and time to GI-3 recovery (toleration of solid food, and flatus or bowel movement) will be secondary endpoints.

Estimated Enrollment = 250, Study Start Date: November 2010, Estimated Study Completion Date: May 2012, Estimated Primary Completion Date: Nov 2011.

ELIGIBILITY:
Inclusion Criteria:

Subject is scheduled to undergo laparoscopic (straight or hand assisted) elective colon resection with primary anastamosis Subject is >18 years of age Subjects can be either male or female Negative pregnancy test (if patient is a premenopausal female) Medically stable as determined by the treating surgeon- i.e., subject has an American Society of Anesthesiologists Physical Status Score of I to III.

Subject understands the study procedures, agrees to participate in the study as per the study protocol, and has voluntarily provided informed consent Patients who will be receiving IV Opioid therapy post surgery for pain management.

Exclusion Criteria:

Subject is pregnant or lactating Subject is currently using opioids or has taken more than 3 doses of opioids (oral or parenteral) in the week prior to surgery.

Subject has complete bowel obstruction Subject is not able to understand the informed consent document or is unable to give informed consent Patients who will receive a thoracic epidural for pain management post surgery. Subject has any medical instability or any condition at screening/enrollment which, in the opinion of the investigator, might confound the results of the study or pose additional risk to the subject during the administration of study procedures.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2010-11; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
length of stay in days | 7-10 days s/p discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Hartford Hospital, Hartford, Connecticut, United States